CLINICAL TRIAL: NCT00320671
Title: Preventing Morbidity in First Episode Schizophrenia, Part II
Brief Title: Comparison of Aripiprazole and Risperidone for the Treatment of People With First-Episode Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Delbert Robinson, Professor of Psychiatry and Molecular Medicine, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH060004-02 (NIH); R01MH060004-02 (NIH)
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: First-episode; Schizoaffective Disorder; Schizophreniform Disorder; Psychotic Disorder Not Otherwise Specified NOS; Aripiprazole; Clozapine; Risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Participants will take aripiprazole (Experimental): Participants will take aripiprazole
  Interventions: Drug: Aripiprazole
- Participants will take risperidone (Experimental): Participants will take risperidone
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Aripiprazole — The dosage for aripiprazole will be 5 mg to 30 mg per day in capsule form. The dose of aripiprazole will be based on the participant's clinical improvement and side effects, which will be evaluated weekly for the first 4 weeks and then every 2 weeks until the 12th week and then monthly until study end.
  Other Names: Abilify
  Arms: Participants will take aripiprazole
Drug: Risperidone — The dosage for risperidone will be 1 mg to 6 mg per day in capsule form. The dose of risperidone will be based on the participant's clinical improvement and side effects, which will be evaluated weekly for the first 4 weeks, then every 2 weeks until the 12th week, and then monthly until the study end.
  Other Names: Risperdal
  Arms: Participants will take risperidone

SUMMARY:
This 52 week long study evaluates the effectiveness of aripiprazole versus risperidone in treating people with first-episode schizophrenia. Patients who do not improve with these medications receive clozapine as their third medication trial.

DETAILED DESCRIPTION:
Schizophrenia is a severely disabling brain disorder. People with schizophrenia often experience hallucinations, delusions, thought disorders, and movement disorders. Medications are available to alleviate the symptoms of schizophrenia, but many cause undesirable side effects. For example, two early second generation antipsychotics, olanzapine and risperidone, have been shown to be effective in treating schizophrenia symptoms, but cause rapid, substantial weight gain. There is a lower risk of such side effects with newer second generation antipsychotics, such as aripiprazole. Little is known, however, about the effectiveness of these newer medications in treating people with first-episode schizophrenia. This study will evaluate the effectiveness of aripiprazole versus risperidone for the treatment of first-episode schizophrenia.

Participants in this double-blind study will be randomly assigned to receive either aripiprazole or risperidone for 12 weeks. Subjects who do not meet response criteria will be continued on their initial blinded antipsychotic for an additional 4 weeks for a total length of 16 weeks of treatment. Subjects who meet response criteria by week 16 will continue on their successful blinded medication for their remaining time in study. Patients who do not respond will be treated with the other medication (aripiprazole or risperidone) that they did not receive during the first 16 weeks of the study. The second antipsychotic trial will last 16 weeks. Patients who respond during the switch phase will be continued on their successful medication during their remaining time in the study. Patients who do not respond to the second medication trial will then be treated with open-label clozapine for 20 weeks. Safety monitoring for clozapine-treated subjects will follow the established procedures for multi-episode patients (e.g . weekly complete blood count (CBC) monitoring). The total length of patient participation is 52 weeks.

During the longitudinal follow-up phase, subjects may be prescribed open-label sodium valproate for manic symptoms and open-label sertraline for symptoms of depression or anxiety empirically responsive to (Selective serotonin reuptake inhibitor)SSRI treatment. Additionally, all participants will take part in a Healthy Lifestyles program aimed at preventing weight gain. The Healthy Lifestyles program will provide psycho-education, supportive psychotherapy, and medication adherence counseling. At each visit, treatment and metabolic outcomes will be assessed. Participants will meet with both a psychiatrist, who will evaluate progress and medication dosage, and a social worker, who will administer the Healthy Lifestyles Program. Upon completion of the study, participants will receive follow-up care from clinical staff members who were not part of the research team.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00000374

ELIGIBILITY:
Inclusion Criteria:

* Current Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, or similar psychotic disorder not otherwise specified, as assessed using the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I/P)
* History of previous antipsychotic medication treatment for a duration of 2 weeks or less
* Current positive symptoms rated 4 (moderate) or more on one or more of the following Brief Psychiatric Rating Scale (BPRS-A) items: conceptual disorganization; grandiosity; hallucinatory behavior; or unusual thought content
* Agrees to use an effective form of contraception

Exclusion Criteria:

* Any serious neurological or endocrine disorder, or any medical condition or treatment known to affect the brain
* Any current medical condition that requires treatment with a medication with psychotropic effects
* At significant risk for suicidal or homicidal behavior
* Cognitive or language limitations, or any other factor that would interfere with a participant's ability to provide informed consent or safely participate in study procedures
* Diagnosis of diabetes, defined as a fasting plasma glucose level of at least 126 mg/dL, or metabolic syndrome, defined as three or more of the following: high blood pressure (greater than 135/85 mmHg); truncal obesity (having a waist circumference greater than 40 inches for men and greater than 35 inches for women); elevated fasting glucose (greater than 110 mg/dL); low HDL-cholesterol (less than 40 mg/dL for men and less than 50 mg/dL for women); or elevated triglycerides (defined as greater than 150 mg/dL)
* Requires treatment with an antidepressant or mood stabilizing medication
* Meets DSM-IV criteria for a current substance-induced psychotic disorder, a psychotic disorder due to a general medical condition, delusional disorder, brief psychotic disorder, shared psychotic disorder, or a mood disorder (major depression or bipolar) with psychotic features
* Any medical conditions that would make treatment with risperidone or aripiprazole medically inadvisable

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Actual)
Dates: Start 2005-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delbert Robinson, MD, Principal Investigator — The North Shore-Long Island Jewish Health System
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Robinson DG, Gallego JA, John M, Petrides G, Hassoun Y, Zhang JP, Lopez L, Braga RJ, Sevy SM, Addington J, Kellner CH, Tohen M, Naraine M, Bennett N, Greenberg J, Lencz T, Correll CU, Kane JM, Malhotra AK. A Randomized Comparison of Aripiprazole and Risperidone for the Acute Treatment of First-Episode Schizophrenia and Related Disorders: 3-Month Outcomes. Schizophr Bull. 2015 Nov;41(6):1227-36. doi: 10.1093/schbul/sbv125. Epub 2015 Sep 3. PMID 26338693

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Will Take Aripiprazole Arm 1: -102 were allocated to Arm 1.
- Participants Will Take Risperidone Arm 2: -96 participants were randomized to to Arm 2
Period: Overall Study
Arm/Group | Participants Will Take Aripiprazole Arm 1 | Participants Will Take Risperidone Arm 2
Started | 102 | 96
Completed | 69 | 58
Not Completed | 33 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Will Take Aripiprazole | Participants Will Take Risperidone | Total
Number analyzed (Participants) | 102 | 96 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 28 | 56
  Between 18 and 65 years | 74 | 68 | 142
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 73 | 70 | 143
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 38 | 35 | 73
  Asian | 22 | 17 | 39
  Caucasian | 21 | 27 | 48
  Hispanic | 11 | 9 | 20
  Other/Mixed | 9 | 7 | 16
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 102 | 96 | 198
Structured Clinical Interview for DSM-IV Axis I Disorders [Number; unit: participants]
  psychosis NOS | 6 | 11 | 17
  Schizoaffective Disorder | 2 | 4 | 6
  Schizophrenia | 72 | 59 | 131
  Schizophreniform Disorder | 22 | 22 | 44
BPRS-A [Mean (Full Range); unit: units on a scale] — Brief Psychiatric Rating Scale-Anchored (BPRS-A) 4 items on this scale were examined to determine subjects responder status: Items 4. Conceptual Disorganization 8. Grandiosity 12. Hallucinations and 15. Unusual Thought Content.
  Only subjects who responded with a 4 or greater on one at least one of theses items were eligible to participate in the study. The scores can range from 0-28 with 28 being the most psychotic and 0 being absolutely no signs of psychosis.
  units on a scale | 14.66 [4 to 28] | 14.42 [4 to 28] | 14.54 [4 to 28]
Scale for the Assessment of Negative [Mean (Standard Deviation); unit: units on a scale] — The Scale for the Assessment of Negative Symptoms (SANS) This scale has 4 subscales Affective flattening, Alogia, Avolition Apathy, and Asociality-anhedonia. Score on these subscales range from 1 normal to 5 severe
  units on a scale
    Affective flattening | 1.85 (0.09) | 1.74 (.09) | 1.795 (.09)
    Alogia | 2.08 (.08) | 1.96 (.09) | 2.02 (.85)
    avolition-apathy | 2.16 (.10) | 2.02 (.10) | 2.09 (.10)
    asociality-anhedonia | 2.19 (.08) | 2.07 (.09) | 2.12 (.85)
Metabolic Outcomes [Least Squares Mean (Standard Deviation); unit: mg/dl]
  Total Cholesterol Baseline | 158.25 (3.15) | 157.01 (3.30) | 157.63 (3.225)
  LDL cholesterol Baseline | 86.37 (2.60) | 88.25 (2.77) | 87.31 (2.685)
  HDL Cholesterol baseline | 55.99 (1.37) | 53.23 (1.40) | 54.61 (1.385)
  Triglycerides baseline | 80.00 (4.48) | 77.41 (4.50) | 78.705 (4.49)
  Fasting glucose baseline | 85.06 (0.69) | 84.60 (0.89) | 84.83 (.79)
hollingshead- index of social position [Mean (Standard Deviation); unit: units on a scale] — The Hollingshead is designed to measure social status of an individual based on educational and occupation. Scores for educational status range from 1 (Grad/Professional School) to a score of 7 ( < than 7 yrs of formal education). For occupation scores range from 1 (high execs, major professionals) to 7 (unskilled employees). Social class scores are obtained for subjects and their self-reported head of household.
  Social Status is based on the formula (Occupation score x 7)+(Education score x 4)-The lower the # the > the social status. Social status scores range from 11 to 77.
  units on a scale
    Highest Educational Level | 4.0 (1.4) | 3.8 (1.1) | 3.9 (1.2)
    Social Class for subject | 4.2 (.8) | 4.6 (3.4) | 4.4 (2.5)
    social class for parent | 3.3 (1.3) | 3.5 (3.6) | 3.4 (2.7)
Marital Status [Number; unit: participants]
  Never Married | 92 | 90 | 182
  Married | 1 | 3 | 4
  Remarried | 1 | 0 | 1
  Divorced | 6 | 3 | 9
  Unknown | 2 | 0 | 2
Fasting insulin [Least Squares Mean (Standard Deviation); unit: uU/ml] | 12.39 (1.10) | 13.10 (1.38) | 12.745 (1.24)
Prolactin Level Female [Least Squares Mean (Standard Deviation); unit: ng/ml] — The measure of dispersion selected is standard deviation; however, the actual number entered below is the STANDARD ERROR.
  ng/ml | 61.84 (7.61) | 65.52 (12.88) | 63.68 (10.24)
Prolactin Level Male [Least Squares Mean (Standard Deviation); unit: ng/ml] — The measure of dispersion selected is standard deviation; however, the actual number entered below is the STANDARD ERROR
  ng/ml | 28.72 (3.05) | 31.50 (3.24) | 30.11 (3.145)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Responded to Treatment
Description: Brief Psychiatric Rating Scale-Anchored (BPRS-A) 4 items on this scale were examined to determine subjects responder status: Items 4. Conceptual Disorganization 8. Grandiosity 12. Hallucinations and 15. Unusual Thought Content. Scores range from-7 (not assessed) to 7 (very severe) Subjects with scores of 3 or less on all 4 items for 2 consecutive visits are deemed responders, subjects with 4 or greater and any of the aforementioned items for 2 consecutive study visits are non responders. Additionally, the subjects response on the Clinical Global Impressions Scale. A Clinical Global Improvement CGI) rating of much or very much improved on 2 consecutive ratings were deemed a responder. Percentages and confidence intervals were used to report response outcome. Response status was assessed throughout the duration of the study; a participant can be deemed a responder any time between weeks 1-week 12. The possible range for this outcome is a score of 4 to 28
Time Frame: this outcome was assessed throughout the study.
Population: BPRS-A and CGI scores for each group were analysed to determine the percentage of participants that responded to apriprazole and risperidone. The threshold for significance was p=.05
Measure: Number (95% Confidence Interval); unit: percentage of response
Groups:
- Percentage of Participants That Reposonded to Aripiprazole: Aripiprazole: The dosage for aripiprazole will be 5 mg to 30 mg per day in capsule form. The dose of aripiprazole will be based on the participant's clinical improvement and side effects, which will be evaluated weekly for the first 4 weeks and then every 2 weeks until the 12th week and then monthly until study end.
- Percentage of Participants That Reposonded to Risperidone: Risperidone: The dosage for risperidone will be 1 mg to 6 mg per day in capsule form. The dose of risperidone will be based on the participant's clinical improvement and side effects, which will be evaluated weekly for the first 4 weeks, then every 2 weeks until the 12th week, and then monthly until the study end.
Arm/Group | Percentage of Participants That Reposonded to Aripiprazole | Percentage of Participants That Reposonded to Risperidone
Number analyzed (Participants) | 102 | 96
percentage of response | 62.8 [50.8 to 74.8] | 56.8 [43.9 to 69.9]
Statistical Analysis 1: Comparison: Percentage of Participants That Reposonded to Risperidone; Test type: Non-Inferiority or Equivalence — Equivalence Analysis; p = .61, Log Rank; Cumulative Response Rates = 56.8, 95% CI 2-sided [43.9 to 69.9] — Only the subjects taking risperidone were analysed in this section
Statistical Analysis 2: Comparison: Percentage of Participants That Reposonded to Aripiprazole; Test type: Non-Inferiority or Equivalence — Equivalence Analysis; p = .61, Log Rank; Cumulative Response Rates = 62.8, 95% CI 2-sided [50.8 to 74.8] — Only subjects taking aripiprazole were analysed in this section

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the duration of the study., up to 12 weeks. The only serious adverse event that was reported was subjects being admitted to the hospital. No other serious adverse occurred throughout the duration of the study.
Arm/Group | Participants Will Take Aripiprazole | Participants Will Take Risperidone
Serious Adverse Events (participants affected / at risk) | 7/102 | 12/96
Other Adverse Events (participants affected / at risk) | 0/102 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Will Take Aripiprazole (N=102) | Participants Will Take Risperidone (N=96)
hospitalization (Psychiatric disorders) | 7 (7) | 12 (12) — subjects were admitted to the hospital

LIMITATIONS AND CAVEATS:
Metabolic data only capture initial effects and may been impacted by Healthy Lifestyles program neg symptoms are only assessed in the initial context of pos symptoms and may not generalize to neg symptoms in the absence of pos symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No